CLINICAL TRIAL: NCT00061087
Title: Treatment of Adult ADHD in Methadone Patients
Brief Title: Treatment of Adult Attention Deficit Hyperactivity Disorder (ADHD) in Methadone Patients - 1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-011444-1,#4184R; R01DA011444 (NIH); 4184R (Other: NYSPI IRB)
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: ADHD; Opioid-Related Disorders; Cocaine Dependence
Keywords: ADHD; Cocaine; Treatment; Methadone
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Opioid-Related Disorders; Cocaine-Related Disorders | interventions — Methylphenidate; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- METHYLPHENIDATE (Active Comparator): Methylphenidate
  Interventions: Drug: Methylphenidate
- BUPROPION (Active Comparator): Bupropion
  Interventions: Drug: Bupropion
- PLACEBO (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate 80mg/day
  Arms: METHYLPHENIDATE
Drug: Bupropion — Bupropion 400mg/day
  Arms: BUPROPION
Other: Placebo — Placebo
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to treat Adult Attention Deficit Hyperactivity Disorder (ADHD) in methadone patients.

DETAILED DESCRIPTION:
This project is a three armed double-blind, placebo-controlled, randomized trial comparing the efficacy of MPH and BPR, relative to each other and to placebo, for treating persistent ADHD in methadone-maintained patients. One hundred and twenty subjects, will be randomized to receive either MPH, BPR, or placebo with equal probability. Randomization will be stratified by site, and whether or not cocaine is also being used. Efficacy will be measured by treatment retention, reduction in illicit drug use and drug craving, improvement of ADHD symptoms and overall functional status.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who meet DSM-IV criteria for opiate dependence and are currently maintained on methadone
* Patients must meet DSM-IV criteria for persistent adult ADHD
* Must be on stable methadone dose for at least 3 weeks
* Individuals positive for HIV will not be excluded.

Exclusion Criteria:

* Patients meeting DSM-IV criteria for current psychiatric disorders (other than ADHD or substance abuse) which requires psychiatric intervention
* Patients who are physiologically dependent on either sedatives or alcohol such that they experience symptoms requiring medical attention during periods of abstinence or significant reduction in amount of use
* Individuals diagnosed with other forms of adult ADHD other than persistent, particularly substance-induced ADHD
* Those who have an unstable medical condition which might make participation hazardous, including but not restricted to: uncontrolled hypertension, (SBP >160, DBP>100, PULSE >110), uncontrolled liver disease, uncontrolled diabetes, acute hepatitis, uncontrolled heart disease as indicated by history or abnormal ECG, glaucoma, or history of urinary retention or seizures, or advanced AIDS will not be included
* Patients who are taking prescription psychotropic medications other than methadone
* Patients who have exhibited suicidal or homicidal behavior within the past two years
* Patients with known sensitivity to MPH or BPR
* Patients with cognitive impairment or who cannot read or understand the self-report assessment forms unaided or are so severely disabled they cannot comply with the requirements of the study.
* Patients unable to give full and informed consent
* Patients with a history of an eating disorder
* Patients recently convicted of a violent crime. (last two years)
* Nursing mothers and pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 1998-02; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Cocaine use based on urine toxicology | collected 3 times per week for 12 weeks of the trial or length of study participation
ADHD symptom severity based on the ADHD Rating scale score | measured once per week for 12 weeks or length of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- Research Foundation for Mental Hygiene, Inc., New York, New York, United States

REFERENCES:
- [Background] Brooks DJ, Vosburg SK, Evans SM, Levin FR. Assessment of cognitive functioning of methadone-maintenance patients: impact of adult ADHD and current cocaine dependence. J Addict Dis. 2006;25(4):15-25. doi: 10.1300/J069v25n04_02. PMID 17088222
- [Result] Levin FR, Evans SM, Brooks DJ, Kalbag AS, Garawi F, Nunes EV. Treatment of methadone-maintained patients with adult ADHD: double-blind comparison of methylphenidate, bupropion and placebo. Drug Alcohol Depend. 2006 Feb 1;81(2):137-48. doi: 10.1016/j.drugalcdep.2005.06.012. Epub 2005 Aug 15. PMID 16102908
- See also: Substance and Research Service of the Division on Substance Abuse of the NYSPI — http://stars.columbia.edu/